CLINICAL TRIAL: NCT02680548
Title: A Pilot Randomized Controlled Trial of Efficacy of Perineural Local Anesthetics and Steroids for Chronic Post-traumatic Neuropathic Pain in the Ankle and the Foot: The PREPLAN Study
Brief Title: Pilot RCT of Efficacy of Perineural Local Anesthetics and Steroids for Chronic Post-traumatic Ankle and Foot Pain
Acronym: PREPLANS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Anuj Bhatia, Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-9584-A
Record Dates: First submitted 2015-12-11; First posted 2016-02-11 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: CHRONIC POST-TRAUMATIC NEUROPATHIC PAIN IN ANKLE AND FOOT
Keywords: ankle pain; foot pain; methylprednisolone; neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Saline Solution; Fluoridation; Bupivacaine; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.9% saline (salt water) (Active Comparator): 0.5mL 0.25% bupivacaine subcutaneous injection, 2-6cc 0.9% saline injection per nerve (20cc max)
  Interventions: Drug: 0.9% saline
- local anesthetic (freezing) (Active Comparator): 0.5mL 0.25% bupivacaine subcutaneous injection, 2-6cc 0.25% bupivacaine per nerve (20cc max)
  Interventions: Drug: 0.25% bupivacaine hydrochloride injectable suspension USP
- local anesthetic (freezing) and steroid (Active Comparator): 0.5mL 0.25% bupivacaine subcutaneous injection, 2-6cc 0.25% bupivacaine and 4mg/cc methylprednisolone per nerve (20cc max)
  Interventions: Drug: 0.25% bupivacaine hydrochloride injectable suspension USP; Drug: 4mg/cc methylprednisolone acetate injectable suspension USP

INTERVENTIONS:
Drug: 0.9% saline
  Other Names: Salt Water
  Arms: 0.9% saline (salt water)
Drug: 0.25% bupivacaine hydrochloride injectable suspension USP
  Other Names: Marcaine
  Arms: local anesthetic (freezing); local anesthetic (freezing) and steroid
Drug: 4mg/cc methylprednisolone acetate injectable suspension USP
  Other Names: Depo-Medrol
  Arms: local anesthetic (freezing) and steroid

SUMMARY:
Injections of local anesthetics (freezing) and steroids are often performed around injured nerves in individuals with nerve injury-related pain. The current standard of medical care is to inject a combination of local anesthetics and steroids around injured nerves, but there is no proof that this is better than injecting only local anesthetic, or even just sterile salt water. There is evidence to believe that injection of local anesthetic (without the steroid) can calm the injured nerve, and provide pain relief from a few days up to a few months. Injection of sterile salt water also has the potential to provide pain relief by breaking scar tissue around the nerve, thereby relieving compression. The aim of this study is to compare pain relief and possible adverse effects from these three different treatments for foot and ankle nerve pain relief.

All 30 participants will be recruited over 9 months from the Altum Health clinic at Toronto Western Hospital. 10 participants will be randomly assigned to each treatment. Each patient will receive 3 injections over 3 weeks or so. Participants will have an in-clinic follow-up at 1 month after the last injection, and a phone follow-up 3 months after the last injection.

This is a small-scale study, and information obtained from this study will help in planning and conduct of a larger study with more participants. The larger study will help determine the best possible option for injection in patients with nerve-related injury pain.

ELIGIBILITY:
Inclusion Criteria:

1. Pain in foot in neuro-anatomically congruent location following trauma (including surgery) for more than three months
2. Physician-reported DN4 scoring confirming neuropathic pain (score > 3/10)
3. Average intensity of pain more than 3/10 on numerical rating score
4. Failed trial of appropriate doses of first line medications for neuropathic pain (anticonvulsants and/or antidepressants) for six weeks

Exclusion Criteria:

1. Age < 18 or age ≥ 80 years
2. Perineural or intra-articular steroid injections in the last 6 months
3. Allergy to local anesthetics and/or steroids
4. Ongoing litigation issues related to the patient's pain
5. Pregnancy
6. Coagulopathy or systemic infection
7. Peripheral neuropathy or myopathy, central neuropathic pain (e.g. post-stroke pain)
8. Infection in the ankle or foot
9. An unstable medical or psychiatric condition
10. Significant catastrophizing as indicated by pain catastrophizing scale (PCS) score equal to or more than 30/52

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Enrollment and retention of participants (SEE DESCRIPTION) | At end of study (1 year)
  Factors considered in assessment: Enrolling at least 75% of eligible patients, enrolling at least 9 patients monthly, retention till study end of at least 90% of participants

SECONDARY OUTCOMES:
Central tendency (mean) and spread (standard deviation) of Numerical Rating Score (NRS) ratings of Foot and Ankle pain | At 1-month and 3-months post-intervention
Change in scores of Pain Catastrophizing Score (PCS) | Baseline and at 1-month post-intervention
Change in scores of Dolores Neuropathique (DN4) | Baseline and at 1-month post-intervention
Change in scores of Neuropathic Pain Symptom Inventory (NPSI) | Baseline and at 1-month post-intervention
Change in scores of anxiety component scores on the Hospital Anxiety and Depression Scale (HADS) | Baseline and at 1-month post-intervention
Change in scores of depression scores on the Patient Health Questionnaire-9 (PHQ-9) | Baseline and at 1-month post-intervention
Change in scores of Brief Pain Inventory interference with activities (BPI-I) | Baseline and at 1-month post-intervention
Change in scores of Short Form-12 (SF-12) | Baseline and at 1-month post-intervention
Change in scores of Lower Extremity Function Score (LEFS) | Baseline and at 1-month post-intervention
Evaluate the impact of study interventions on requirement for opioids (measured as average daily oral morphine equivalents in mg) and neuropathic medications (average daily doses of gabapentin and/or amitriptyline in mg) | At end of study (1 year)
Change in pre- and post-intervention levels of blood glucose and blood pressure | Baseline and at 1-month post-intervention
Measure incidence of infections at the injection site, skin discoloration or atrophy at the injection site, fractures, and evidence of myopathy | Baseline and at 1-month post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Bhatia, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatia A, Bril V, Brull RT, Perruccio A, Wijeysundera D, Alvi S, Lau J, Gandhi R, Mahomed N, Davis AM. Study protocol for a pilot, randomised, double-blinded, placebo controlled trial of perineural local anaesthetics and steroids for chronic post-traumatic neuropathic pain in the ankle and foot: the PREPLANS study. BMJ Open. 2016 Jun 22;6(6):e012293. doi: 10.1136/bmjopen-2016-012293. PMID 27334885